CLINICAL TRIAL: NCT05080270
Title: Feasibility Study of Tolerogenic Fibroblasts in Patients With Refractory Multiple Sclerosis
Acronym: MSFibroblast
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: FibroBiologics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fibroblast_MS_safety2021
Record Dates: First submitted 2021-10-05; First posted 2021-10-15 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis
Keywords: MS; Cell Therapy; Fibroblasts; Fibrobiologics; Stem cells; regenerative medicine; tissue regeneration; Immune modulation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The proposed study will assess primary safety and secondary efficacy endpoints of allogeneic tolerogenic fibroblasts administered through Intravenous infusion at a single dose of 100 million cells to 5 patients with relapsing remitting MS resistant to interferon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tolerogenic fibroblasts administered via intravenous infusion (Experimental): A single dose of 100 million tolerogenic fibroblasts administered via intravenous infusion.
  Interventions: Biological: Tolerogenic Fibroblasts

INTERVENTIONS:
Biological: Tolerogenic Fibroblasts — administrating single dose of 100 million tolerogenic fibroblasts via intravenous infusion

SUMMARY:
Fibroblasts have demonstrated potent immune modulatory and therapeutic activity in the experimental autoimmune encephalomyelitis (EAE) model of multiple sclerosis, as well as in other models of autoimmune and inflammatory diseases.

This study will assess primary safety and secondary efficacy endpoints of intravenous administration of 100 million tolerogenic fibroblasts to 5 patients with relapsing remitting MS resistant to interferon. While the safety of fibroblasts administered clinically is established, it is unknown whether these cells are effective in the treatment of multiple sclerosis (MS).

Our hypothesis is that the tolerogenic fibroblasts will be well-tolerated and meet our primary objective. In addition, The investigators are optimistic that they will see signs of efficacy based on the following: Neurological assessment of the MS functional composite assessment which comprises of EDSS, the expanded EDSS (Rating Neurologic Impairment in Multiple Sclerosis, the Scripps neurological rating scale (NRS), paced auditory serial addition test (PASAT), the nine-hole peg test, and 25-foot walking time, short-form 36 (SF-36) quality of life questionnaire and gadolinium-enhanced MRI scans of the brain and cervical spinal cord.

DETAILED DESCRIPTION:
Fibroblasts have demonstrated potent immune modulatory and therapeutic activity in the experimental autoimmune encephalomyelitis (EAE) model of multiple sclerosis, as well as in other models of autoimmune and inflammatory diseases. Mechanistically, tolerogenic fibroblasts produce anti-inflammatory and immune modulatory factors, which appear to be therapeutic in the context of autoimmunity, including IL-10 and TGF-beta. Additionally, tolerogenic fibroblasts produce neurotrophic mediators that enhance myelin production and/or prevent neuronal apoptosis.

This study will assess primary safety and secondary efficacy endpoints of intravenous administration of 100 million tolerogenic fibroblasts to 5 patients with relapsing remitting MS resistant to interferon. While the safety of fibroblasts administered clinically is established, it is unknown whether these cells are effective in the treatment of multiple sclerosis (MS).

Research Hypothesis: Intravenous administration of 100 million tolerogenic fibroblasts will be well tolerated and induce a therapeutic effect in relapse remitting MS patients.

Rationale: The family of Mesenchymal Stem Cells (MSCs) is immune-modulatory, and bone marrow MSCs (BM-MSCs) have induced therapeutic responses in patients with MS [1]. Tolerogenic fibroblasts possess superior immune modulatory activity compared to BM-MSCs and adipose MSCs. The investigators, therefore, seek to perform a five-patient trial to assess the safety and signs of efficacy of this cell population in MS patients resistant to interferon.

The trial's primary objective is freedom from treatment-associated adverse events at 1, 2, 4, 8, and 16 weeks post-treatment. The study's secondary objective will be efficacy as assessed at baseline, weeks 2, 4, 8, and 16. The results will be quantified based on the following: Neurological assessment of the MS functional composite assessment, which comprises of EDSS, the expanded EDSS (Rating Neurologic Impairment in Multiple Sclerosis, the Scripps neurological rating scale (NRS), paced auditory serial addition test (PASAT), the nine-hole peg test, and 25-foot walking time, short-form 36 (SF-36) quality of life questionnaire and gadolinium-enhanced MRI scans of the brain and cervical spinal cord.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to sign an informed consent and capable of understanding the features of this clinical trial.
2. Willing to keep a weekly diary and undergo observation for four months
3. Non-pregnant patients 18-55 years of age with MS according to the revised McDonald criteria and meeting the Possner criteria for clinically defined MS.
4. EDSS scores of 2·0 to 5·5 points assessed at least three months after the last acute attack of MS.

Exclusion Criteria:

1. Patients with evidence of active proliferative retinopathy.
2. Patients with poorly controlled diabetes mellitus (HbA1C > 8.5%).
3. Patients with renal insufficiency (Creatinine > 2.5) or failure.
4. Infection as evidenced by WBC count of >15,000 k/cumm and/or temperature >38C.
5. History of organ transplant.
6. History of previous or active malignancy, except for localized cutaneous basal or squamous cell carcinoma or carcinoma in situ of the cervix
7. History of sickle cell anemia
8. Cardiovascular conditions:

   1. Exercise limiting angina ( Canadian Cardiovascular Society Class greater or equal to 3
   2. Congestive heart failure (New York Heart Association class greater or equal to 3
   3. Unstable angina
   4. Acute ST elevation myocardial infarction (MI) within one month
   5. Transient ischemic attack or stroke within one month
   6. Severe valvular disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse even monitoring of subjects for 4 hours after infusion | Monitoring during the Intravenous infusion of allogeneic tolerogenic fibroblasts, and continued for 4 hours after infusion
  Monitor subjects for possible treatment-related acute immune symptoms or vascular occlusion symptoms during the administration of the allogeneic tolerogenic fibroblasts via intravenous infusion.
Safety: Complete Blood Count to monitor inflammation markers | Day before infusion to establish a baseline, week 8, and week 16 after infusion
  Complete Blood Count used to monitor inflammation markers included white blood cell (WBC), neutrophil (N), lymphocyte (L), neutrophil-lymphocyte ratio (NLR), mean platelet volume (MPV), and platelet-lymphocyte ratio. This safety test is to monitor subjects for inflammation during the course of the study, relating to the course of the disease, or allogeneic tolerogenic fibroblasts administered through Intravenous infusion
Safety: Serum chemistry to monitor impact on serum chemistry | Day before infusion to establish a baseline, week 8, and week 16 after infusion
  This test will measure the amount of certain substances in serum samples, including electrolytes (such as sodium, potassium, and chloride), fats, proteins, glucose (sugar), and enzymes. Blood chemistry tests give essential information about how well a person's kidneys, liver, and other organs are working. An abnormal amount of a substance in the blood can be a sign of disease or a side effect of treatment. Blood chemistry tests help diagnose and monitor many conditions before, during, and after treatment. Also called blood chemistry study.
Safety: 12-lead Electrocardiogram (ECG) to monitor cardiovascular health | Day before infusion to establish a baseline, week 8, and week 16 after infusion
  A 12-lead electrocardiogram will be used to monitor the baseline cardiovascular health of the participants and continue to monitor their cardiovascular health during the course of the study measuring heart rate, blood pressure, ventricular rate, PR interval, RP interval, QRS interval, and GT interval. This safety test is to monitor the subjects for cardiac events related to the course of the disease, or allogeneic tolerogenic fibroblasts administered through Intravenous infusion

SECONDARY OUTCOMES:
Efficacy: Expanded Disability Status Scale (EDSS) to quantify disability scale and monitors changes | Day before infusion to establish a baseline, week 8, and week 16 after infusion
  The Expanded Disability Status Scale (EDSS) quantifies disability in multiple sclerosis and monitors changes in the level of disability over time. The test is based on neurological examination and impact on Functional Systems representing network of neurons in the brain. It is widely used in clinical trials and the assessment of people with MS. The scale was developed by a neurologist called John Kurtzke in 1983 as an advance from his previous 10 step Disability Status Scale (DSS). The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Efficacy: Paced Auditory Serial Addition Test (PASAT) to measure cognitive function and processing speed | Day before infusion to establish a baseline, week 8, and week 16 after infusion
  PASAT is a measure of cognitive function that assesses auditory information processing speed, flexibility, and calculation ability. The test was developed by Gronwell in 1977 and later adapted by Rao and colleagues in 1989 for use in MS. The PASAT is presented using audio cassette tape or compact disk to ensure standardization in the rate of stimulus presentation. In the test, single digits are presented every 3 seconds, and the patient must add each new digit to the one immediately prior to it. Shorter inter-stimulus intervals, e.g., 2 seconds or less, have also been used with the PASAT but tend to increase the difficulty of the task.
Efficacy: Nine-Hole Peg Test to measure and quantify upper extermity function | Day before infusion to establish a baseline, week 8, and week 16 after infusion
  The 9-HPT is a brief, standardized, quantitative test of upper extremity function. Both the dominant and non-dominant hands are tested twice. The patient is seated at a table with a small, shallow container holding nine pegs and a wood or plastic block containing nine empty holes. On a start command when a stopwatch is started, the patient picks up the nine pegs one at a time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand.
Efficacy: Timed 25-Foot Walk Test to quantify mobility and leg function | Day before infusion to establish a baseline, week 8, and week 16 after infusion
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.
Efficacy: Gadolinium Enhanced MRI to detect demyelinated areas of the nerves | Day before infusion to establish a baseline, and week 16 after infusion
  Gadolinium Enhanced MRI is used to detect demyelinated areas of the nerves in the brain and cervical spinal cord. These Damaged areas can be observed by MRI presented as plaques, and the intensity of the plaques can determine the age of multiple sclerosis caused lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Khoja, Ph.D., Study Director — FibroBiologics
Locations (1):
- Servicios Medicos UCC, S.C., Tijuana, Estado de Baja California, Mexico

REFERENCES:
- [Background] Connick P, Kolappan M, Crawley C, Webber DJ, Patani R, Michell AW, Du MQ, Luan SL, Altmann DR, Thompson AJ, Compston A, Scott MA, Miller DH, Chandran S. Autologous mesenchymal stem cells for the treatment of secondary progressive multiple sclerosis: an open-label phase 2a proof-of-concept study. Lancet Neurol. 2012 Feb;11(2):150-6. doi: 10.1016/S1474-4422(11)70305-2. Epub 2012 Jan 10. PMID 22236384
- [Background] Kantarci O, Wingerchuk D. Epidemiology and natural history of multiple sclerosis: new insights. Curr Opin Neurol. 2006 Jun;19(3):248-54. doi: 10.1097/01.wco.0000227033.47458.82. PMID 16702830
- [Background] Evans C, Beland SG, Kulaga S, Wolfson C, Kingwell E, Marriott J, Koch M, Makhani N, Morrow S, Fisk J, Dykeman J, Jette N, Pringsheim T, Marrie RA. Incidence and prevalence of multiple sclerosis in the Americas: a systematic review. Neuroepidemiology. 2013;40(3):195-210. doi: 10.1159/000342779. Epub 2013 Jan 24. PMID 23363936
- [Background] Ghasemi N, Razavi S, Nikzad E. Multiple Sclerosis: Pathogenesis, Symptoms, Diagnoses and Cell-Based Therapy. Cell J. 2017 Apr-Jun;19(1):1-10. doi: 10.22074/cellj.2016.4867. Epub 2016 Dec 21. PMID 28367411
- [Background] Navikas V, Link H. Review: cytokines and the pathogenesis of multiple sclerosis. J Neurosci Res. 1996 Aug 15;45(4):322-33. doi: 10.1002/(SICI)1097-4547(19960815)45:43.0.CO;2-B. PMID 8872892
- [Background] Marrie RA, Elliott L, Marriott J, Cossoy M, Blanchard J, Leung S, Yu N. Effect of comorbidity on mortality in multiple sclerosis. Neurology. 2015 Jul 21;85(3):240-7. doi: 10.1212/WNL.0000000000001718. Epub 2015 May 27. PMID 26019190
- [Background] Goldman MD, Motl RW, Rudick RA. Possible clinical outcome measures for clinical trials in patients with multiple sclerosis. Ther Adv Neurol Disord. 2010 Jul;3(4):229-39. doi: 10.1177/1756285610374117. PMID 21179614
- [Background] SCHUMACHER GA, BEEBE G, KIBLER RF, KURLAND LT, KURTZKE JF, MCDOWELL F, NAGLER B, SIBLEY WA, TOURTELLOTTE WW, WILLMON TL. PROBLEMS OF EXPERIMENTAL TRIALS OF THERAPY IN MULTIPLE SCLEROSIS: REPORT BY THE PANEL ON THE EVALUATION OF EXPERIMENTAL TRIALS OF THERAPY IN MULTIPLE SCLEROSIS. Ann N Y Acad Sci. 1965 Mar 31;122:552-68. doi: 10.1111/j.1749-6632.1965.tb20235.x. No abstract available. PMID 14313512
- [Background] Polman CH, Rudick RA. The multiple sclerosis functional composite: a clinically meaningful measure of disability. Neurology. 2010 Apr 27;74 Suppl 3:S8-15. doi: 10.1212/WNL.0b013e3181dbb571. PMID 20421572
- [Background] Rodgers JM, Robinson AP, Miller SD. Strategies for protecting oligodendrocytes and enhancing remyelination in multiple sclerosis. Discov Med. 2013 Aug;16(86):53-63. PMID 23911232
- [Background] Ernstsson O, Gyllensten H, Alexanderson K, Tinghog P, Friberg E, Norlund A. Cost of Illness of Multiple Sclerosis - A Systematic Review. PLoS One. 2016 Jul 13;11(7):e0159129. doi: 10.1371/journal.pone.0159129. eCollection 2016. PMID 27411042
- [Background] Hartung DM, Bourdette DN, Ahmed SM, Whitham RH. The cost of multiple sclerosis drugs in the US and the pharmaceutical industry: Too big to fail? Neurology. 2015 May 26;84(21):2185-92. doi: 10.1212/WNL.0000000000001608. Epub 2015 Apr 24. PMID 25911108
- [Background] Frampton JE. Ocrelizumab: First Global Approval. Drugs. 2017 Jun;77(9):1035-1041. doi: 10.1007/s40265-017-0757-6. PMID 28523586
- [Background] Offner H, Sinha S, Burrows GG, Ferro AJ, Vandenbark AA. RTL therapy for multiple sclerosis: a Phase I clinical study. J Neuroimmunol. 2011 Feb;231(1-2):7-14. doi: 10.1016/j.jneuroim.2010.09.013. Epub 2010 Oct 20. PMID 20965577
- [Background] Karussis D, Karageorgiou C, Vaknin-Dembinsky A, Gowda-Kurkalli B, Gomori JM, Kassis I, Bulte JW, Petrou P, Ben-Hur T, Abramsky O, Slavin S. Safety and immunological effects of mesenchymal stem cell transplantation in patients with multiple sclerosis and amyotrophic lateral sclerosis. Arch Neurol. 2010 Oct;67(10):1187-94. doi: 10.1001/archneurol.2010.248. PMID 20937945
- [Background] Burton JM, Kimball S, Vieth R, Bar-Or A, Dosch HM, Cheung R, Gagne D, D'Souza C, Ursell M, O'Connor P. A phase I/II dose-escalation trial of vitamin D3 and calcium in multiple sclerosis. Neurology. 2010 Jun 8;74(23):1852-9. doi: 10.1212/WNL.0b013e3181e1cec2. Epub 2010 Apr 28. PMID 20427749
- [Background] Bielekova B, Richert N, Howard T, Packer AN, Blevins G, Ohayon J, McFarland HF, Sturzebecher CS, Martin R. Treatment with the phosphodiesterase type-4 inhibitor rolipram fails to inhibit blood--brain barrier disruption in multiple sclerosis. Mult Scler. 2009 Oct;15(10):1206-14. doi: 10.1177/1352458509345903. Epub 2009 Sep 23. PMID 19776093
- See also: EDSS description — https://mstrust.org.uk/a-z/expanded-disability-status-scale-edss
- See also: Multiple Sclerosis overview — http://emedicine.medscape.com/article/1146199-overview
- See also: Diagnosing Multiple Sclerosis and Evaluating Disease Activity — https://mymsaa.org/ms-information/overview/diagnosing-evaluating/